CLINICAL TRIAL: NCT03110185
Title: Postoperative Delirium: Brain Vulnerability and Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Ben Palanca, Assistant Professor, Washington University School of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 201511004
Record Dates: First submitted 2016-01-14; First posted 2017-04-12 (Actual); Results first posted 2020-06-02 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Delirium; Postoperative Complications
MeSH Terms: conditions — Delirium; Postoperative Complications | interventions — Electroencephalography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- delirium (Other): Patients in the cardiothoracic ICU diagnosed with postoperative delirium. Subjects will wear a diffuse optical tomography device in addition to the normal monitors. A non-contrast functional MRI will be performed.
  Interventions: Device: EEG; Device: fcDOT; Device: fcMRI
- no delirium (Other): Patients in the cardiothoracic ICU not diagnosed with postoperative delirium. Subjects will be monitored in the same way as the delirium arm
  Interventions: Device: EEG; Device: fcDOT; Device: fcMRI

INTERVENTIONS:
Device: EEG — Brain activity will be recorded to evaluate differences in brain activity between patients with a delirium diagnosis and non-delirious control patients.
  Other Names: brain monitoring in delirious postoperative patients
Device: fcDOT — Brain activity will be recorded to evaluate differences in brain activity between patients with a delirium diagnosis and non-delirious control patients.
  Other Names: brain monitoring in delirious postoperative patients
Device: fcMRI — Brain activity will be recorded to evaluate differences in brain activity between patients with a delirium diagnosis and non-delirious control patients.
  Other Names: brain monitoring in delirious postoperative patients

SUMMARY:
In this study, we propose to use EEG and a brain imaging technique known as diffuse optical tomography (DOT) to study when people are in delirium and when they recovery. We plan to also compare brain function of patients who recovered from delirium to patients who did not have delirium using DOT and fMRI. We will also continually monitor the participant's EMR to help coordinate timing of study procedures, as well as to collect information pertaining to their surgery, recovery progress, and indicators of mental status including delirium.

DETAILED DESCRIPTION:
Postoperative delirium - a mental state of confusion, inattention, and impaired thought - is a potentially life-threatening condition. As many as half of patients that have heart and non heart-related surgery will experience postoperative delirium. Patients diagnosed with postoperative delirium have poorer outcomes and longer hospitalizations. Unfortunately, it is an under-diagnosed condition with a variable delay in when it appears. Additionally, there are no objective tools or tests that can be before or after surgery to anticipate and identify those patients who are at risk. Electroencephalography [EEG] and functional magnetic resonance imaging [fMRI] have helped us understand the changes in the brain during delirium. These suggest that a weakening in correlated activity within a group of brain regions, known as the default mode network (DMN), may be related to delirium.

ELIGIBILITY:
Common inclusion criteria:

1. Age ≥ 60
2. Surgery requiring cardiopulmonary bypass (CPB) for coronary artery bypass grafting, septal myectomy and/or heart valve repair/replacement
3. English speaking.

Common exclusion criteria:

1. Implanted pacemaker
2. Automatic internal cardiac defibrillator or other implant for which non-contrast magnetic resonance imaging (MRI) is contraindicated
3. Concomitant aortic or cerebrovascular procedure
4. Inability to lay flat or still for MRI
5. Legal blindness or severe deafness
6. Seizure history
7. Known focal brain lesion larger than 3 cm.

Delirium Case Arm:

1. Delirious as diagnosed by the Confusion Assessment Method (CAM)/ Confusion Assessment Method for the Intensive Care Unit (CAM-ICU) at some point during postoperative day 1-5.

Postoperative Control Arm:

1. Not delirious as diagnosed by the CAM/CAM-ICU on postoperative day 1-5.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2015-11-25 (Actual); Primary Completion 2019-03-08 (Actual); Study Completion 2019-03-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ben Palanca, MD, PhD, MSc, Principal Investigator — Washington University School of Medicine
Locations (1):
- Barnes-Jewish Hospital/Washington University in St. Louis School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were either recruited pre- or post-operatively for study procedures depending on availability of equipment and research staff.
Pre-assignment Details: Participants were not assigned to groups, as baseline delirium status determined which group the participants fell into (delirium vs. no delirium).
Groups:
- Delirium: Patients in the cardiothoracic ICU diagnosed with postoperative delirium. Subjects will wear a diffuse optical tomography device in addition to the normal monitors. A non-contrast functional MRI will be performed.
  fcMRI: Brain activity will be recorded using MRI to evaluate differences in brain activity between patients with a delirium diagnosis and non-delirious control patients.
- No Delirium: Patients in the cardiothoracic ICU not diagnosed with postoperative delirium. Subjects will be monitored in the same way as the delirium arm
  fcMRI: Brain activity will be recorded using MRI to evaluate differences in brain activity between patients with a delirium diagnosis and non-delirious control patients.
Period: Overall Study
Arm/Group | Delirium | No Delirium
Started | 27 | 64
Completed | 17 | 33
Not Completed | 10 | 31
Not completed — Death | 0 | 1
Not completed — Withdrawal by Subject | 2 | 7
Not completed — Time Constraints | 0 | 6
Not completed — Conflict with care | 5 | 12
Not completed — Protocol Violation | 1 | 4
Not completed — MRI Incompatible | 2 | 0
Not completed — Patient Refusal | 0 | 1

BASELINE CHARACTERISTICS:
Population: 9 participants who completed study procedures were excluded from analyses due to poor data quality.
Groups:
- Total: Total of all reporting groups
Arm/Group | Delirium | No Delirium | Total
Number analyzed (Participants) | 13 | 28 | 41
Age, Continuous [Median (Full Range); unit: years] | 74 [61 to 88] | 68.5 [60 to 84] | 70 [60 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 10 | 25 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 13 | 28 | 41
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 12 | 28 | 40
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: EEG During Delirium and After Recovery and in Patient Controls.
Description: Delta (0.5-4 Hz), theta (4-8 Hz), and alpha (8-12 Hz) EEG waveforms.
Time Frame: Data acquisition will occur on 4 separate days between postoperative days 1-8.
Population: Due to time constraints and limited availability of staff and the EEG technology, no participants completed both the pre-operative and post-operative EEG. Therefore, these data were not analyzed.
Groups:
- Delirium: Patients in the cardiothoracic ICU diagnosed with postoperative delirium. Subjects will wear a diffuse optical tomography device in addition to the normal monitors. A non-contrast functional MRI will be performed.
  EEG, fcDOT, fcMRI: Brain activity will be recorded using EEG, fcDOT and MRI to evaluate differences in brain activity between patients with a delirium diagnosis and non-delirious control patients.
- No Delirium: Patients in the cardiothoracic ICU not diagnosed with postoperative delirium. Subjects will be monitored in the same way as the delirium arm
  EEG, fcDOT, fcMRI: Brain activity will be recorded using EEG, fcDOT and MRI to evaluate differences in brain activity between patients with a delirium diagnosis and non-delirious control patients.
Arm/Group | Delirium | No Delirium
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Functional Connectivity Diffuse Optical Tomography (fcDOT) in Patients During Delirium and After Recovery and in Patient Controls
Description: Functional connectivity between anterior and posterior Default Mode Network regions using diffuse optical imaging.
Time Frame: Data acquisition will occur on 4 separate days between postoperative days 1-8.
Population: Due to the limited availability of staff and the DOT equipment, no participants completed both the pre-operative and post-operative DOT. Therefore, these data were not analyzed.
Arm/Group | Delirium | No Delirium
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Functional Connectivity Magnetic Resonance Imaging (fcMRI) in Patients After Recovery From Delirium and in Patient Controls.
Description: Functional connectivity between anterior and posterior Default Mode Network regions assessed from resting-state fcMRI acquired during eyes open wakefulness. Scored using r-value, using a scale of -1 to +1. -1 = strong negative correlation, +1 = strong positive correlation
Time Frame: Within one month after hospital discharge.
Population: Nine participants (4 delirium, and 5 no delirium) who completed study procedures were excluded from analyses due to poor data quality or lack of post-operative delirium data.
Measure: Median (Inter-Quartile Range); unit: r-value
Arm/Group | Delirium | no Delirium
Number analyzed (Participants) | 13 | 28
r-value | 0.1321 [0.008 to 0.2562] | 0.1731 [0.1048 to 0.2414]
Statistical Analysis 1: Comparison: Delirium vs no Delirium; Test type: Other — Correlation; p = 0.0761, Regression, Logistic — Delirium Incidence. There were no multiple comparisons, but includes age as a regressor. a priori threshold was p < 0.05; Generalized logistic regression for delirium incidence and total DMN fc with age as a regressor

ADVERSE EVENTS:
Time Frame: 4 visits over several weeks (up to 3 months)
Arm/Group | Delirium | no Delirium
All-Cause Mortality (participants affected / at risk) | 0/17 | 2/33
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/33
Other Adverse Events (participants affected / at risk) | 0/17 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-26): https://cdn.clinicaltrials.gov/large-docs/85/NCT03110185/Prot_SAP_000.pdf